CLINICAL TRIAL: NCT02436317
Title: Influence of Point of Care Ultrasonography on Outcome of Inpatients Admitted To the Internal Ward
Brief Title: Point of Care Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Yael Ben Baruch Golan MD, Dr. Yael Golan, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: sor12115ctil; SCRC15008 (Other: Soroka CRC)
Record Dates: First submitted 2015-04-21; First posted 2015-05-06 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Abnormalities; Cardiovascular Abnormalities; Hemodynamic Instability
Keywords: Point Of Care Ultrasonography; Soroka University Medical Center; Heart Failure; cardiovascular
MeSH Terms: conditions — Cardiovascular Abnormalities; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): All patients included in intervention group will be examined with an ultrasound machine with cardiac probe and vascular probe [Saote/ Mylab 5/ Italy] using both 2 dimensional and color Doppler imaging modalities according to our local point of care ultrasonography protocol.
  Including demographic and medical data collection. Also, a wellbeing questionnaire will be filled by the investigator.
  Interventions: Device: Point Of Care Ultrasound
- Control group (No Intervention): All patients included in the control group won't be examined with an ultrasound machine. Participation including demographic and medical data collection. Also, a wellbeing questionnaire will be filled by the investigator.

INTERVENTIONS:
Device: Point Of Care Ultrasound — Examination with an ultrasound machine
  Other Names: MyLabfive
  Arms: Study group

SUMMARY:
This is a Prospective, Double-center, randomized clinical trial. The purpose of the trial is to evaluate the benefit of adding POC US to the management of inpatients admitted to the internal ward with respiratory, cardiovascular or hemodynamic abnormalities.

DETAILED DESCRIPTION:
This is a Prospective, Double-center, randomized clinical trial. The purpose of the trial is to evaluate the benefit of adding POC US to the management of inpatients admitted to the internal ward with respiratory, cardiovascular or hemodynamic abnormalities.

This is a stage 1 pilot trial aimed to provide better understanding on the study population and study groups. This trial will comprise a total of 60 patients, 30 subjects on the intervention group and an equal number on the control group. The results of this pilot trial will be to design a larger trial and calculate a required sample size.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to internal ward
2. Age ≥ 18
3. No previous internal ward admission within the last 6 months
4. At least one symptom or sign of the following on admission:

   * Respiratory abnormalities: Dyspnea, RR>20, O2 SAT<90% requirement of oxygen or non-invasive ventilation or mechanical ventilation
   * Cardiovascular abnormalities: Chest pain, HR>100, new/worsening peripheral edema, newly diagnosed ECG changes
   * Hemodynamic instability: SBP<90 mmHg or on vasopressor infusion or pre-renal azotemia

Exclusion Criteria:

1. Patients with cognitive impairment or cannot sign informed consent.
2. Subject enrolled in a different study
3. Patients with end stage disease receiving Palliative/end of life treatments.
4. Pregnant patients.
5. Patients that were given a consult by one of the research members pre enrollment
6. Patient under responsibility of one of the study team members

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07-19 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization | 1 month

SECONDARY OUTCOMES:
Readmission rates | 15 months

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Result] Preston DL, Ron E, Tokuoka S, Funamoto S, Nishi N, Soda M, Mabuchi K, Kodama K. Solid cancer incidence in atomic bomb survivors: 1958-1998. Radiat Res. 2007 Jul;168(1):1-64. doi: 10.1667/RR0763.1. PMID 17722996
- [Result] Pearce MS, Salotti JA, Little MP, McHugh K, Lee C, Kim KP, Howe NL, Ronckers CM, Rajaraman P, Sir Craft AW, Parker L, Berrington de Gonzalez A. Radiation exposure from CT scans in childhood and subsequent risk of leukaemia and brain tumours: a retrospective cohort study. Lancet. 2012 Aug 4;380(9840):499-505. doi: 10.1016/S0140-6736(12)60815-0. Epub 2012 Jun 7. PMID 22681860
- [Result] Moore CL, Copel JA. Point-of-care ultrasonography. N Engl J Med. 2011 Feb 24;364(8):749-57. doi: 10.1056/NEJMra0909487. No abstract available. PMID 21345104
- [Result] Hothi SS, Sprigings D, Chambers J. Point-of-care cardiac ultrasound in acute medicine--the quick scan. Clin Med (Lond). 2014 Dec;14(6):608-11. doi: 10.7861/clinmedicine.14-6-608. PMID 25468845
- [Result] Labovitz AJ, Noble VE, Bierig M, Goldstein SA, Jones R, Kort S, Porter TR, Spencer KT, Tayal VS, Wei K. Focused cardiac ultrasound in the emergent setting: a consensus statement of the American Society of Echocardiography and American College of Emergency Physicians. J Am Soc Echocardiogr. 2010 Dec;23(12):1225-30. doi: 10.1016/j.echo.2010.10.005. PMID 21111923
- [Result] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Result] Oren-Grinberg A, Talmor D, Brown SM. Focused critical care echocardiography. Crit Care Med. 2013 Nov;41(11):2618-26. doi: 10.1097/CCM.0b013e31829e4dc5. PMID 23989172
- [Result] Kobal SL, Atar S, Siegel RJ. Hand-carried ultrasound improves the bedside cardiovascular examination. Chest. 2004 Sep;126(3):693-701. doi: 10.1378/chest.126.3.693. PMID 15364744
- [Result] Spencer KT, Anderson AS, Bhargava A, Bales AC, Sorrentino M, Furlong K, Lang RM. Physician-performed point-of-care echocardiography using a laptop platform compared with physical examination in the cardiovascular patient. J Am Coll Cardiol. 2001 Jun 15;37(8):2013-8. doi: 10.1016/s0735-1097(01)01288-8. PMID 11419879
- [Result] Lichtenstein D, Goldstein I, Mourgeon E, Cluzel P, Grenier P, Rouby JJ. Comparative diagnostic performances of auscultation, chest radiography, and lung ultrasonography in acute respiratory distress syndrome. Anesthesiology. 2004 Jan;100(1):9-15. doi: 10.1097/00000542-200401000-00006. PMID 14695718
- [Result] Mjolstad OC, Dalen H, Graven T, Kleinau JO, Salvesen O, Haugen BO. Routinely adding ultrasound examinations by pocket-sized ultrasound devices improves inpatient diagnostics in a medical department. Eur J Intern Med. 2012 Mar;23(2):185-91. doi: 10.1016/j.ejim.2011.10.009. Epub 2011 Nov 9. PMID 22284252
- [Result] Laursen CB, Sloth E, Lassen AT, Christensen Rd, Lambrechtsen J, Madsen PH, Henriksen DP, Davidsen JR, Rasmussen F. Point-of-care ultrasonography in patients admitted with respiratory symptoms: a single-blind, randomised controlled trial. Lancet Respir Med. 2014 Aug;2(8):638-46. doi: 10.1016/S2213-2600(14)70135-3. Epub 2014 Jul 3. PMID 24998674
- [Result] Al Deeb M, Barbic S, Featherstone R, Dankoff J, Barbic D. Point-of-care ultrasonography for the diagnosis of acute cardiogenic pulmonary edema in patients presenting with acute dyspnea: a systematic review and meta-analysis. Acad Emerg Med. 2014 Aug;21(8):843-52. doi: 10.1111/acem.12435. PMID 25176151
- [Result] Fedson S, Neithardt G, Thomas P, Lickerman A, Radzienda M, DeCara JM, Lang RM, Spencer KT. Unsuspected clinically important findings detected with a small portable ultrasound device in patients admitted to a general medicine service. J Am Soc Echocardiogr. 2003 Sep;16(9):901-5. doi: 10.1016/S0894-7317(03)00426-7. PMID 12931101
- [Result] Laursen CB, Sloth E, Lambrechtsen J, Lassen AT, Madsen PH, Henriksen DP, Davidsen JR, Rasmussen F. Focused sonography of the heart, lungs, and deep veins identifies missed life-threatening conditions in admitted patients with acute respiratory symptoms. Chest. 2013 Dec;144(6):1868-1875. doi: 10.1378/chest.13-0882. PMID 23948720
- [Result] Thiel SW, Kollef MH, Isakow W. Non-invasive stroke volume measurement and passive leg raising predict volume responsiveness in medical ICU patients: an observational cohort study. Crit Care. 2009;13(4):R111. doi: 10.1186/cc7955. Epub 2009 Jul 8. PMID 19586543